CLINICAL TRIAL: NCT02681653
Title: Prospective Randomized Study to Assess Impact of Statins in Septic Shock
Brief Title: Study the Impact of Statins in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/IMP/IEC/56/19.08.2011
Record Dates: First submitted 2015-09-15; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2015-12

CONDITIONS: Septic Shock
Keywords: Statins; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin (Active Comparator): Atorvastatin, 40 mg for 7 days in patients of septic shock admitted to ICU
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Matched placebo, 40 mg for 7 days in patients of septic shock admitted to ICU
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin or placebo given for 7 days to patients of septic shock admitted to ICU
  Arms: Statin
Drug: Placebo — Equally matched placebo for 7 days to patients of septic shock admitted to ICU
  Arms: Placebo

SUMMARY:
Sepsis is a common, expensive, frequently fatal and highly complex inflammatory syndrome wherein multiple cellular and humoral pathways are involved. Since it's a multifactorial syndrome merely blocking one of the various inflammatory pathways may not suffice to provide effective treatment and this may partly explain why most of the adjunctive therapies developed for severe sepsis have yielded disappointing results in rigorous clinical trials. Statins have varied pleiotropic effects on the inflammatory mediators and there addition to the current adjuvant therapies in septic shock may help in reduction of mortality. The present trial aims to study survival benefit and changes in bio-marker levels in septic shock.

Adult patients (>=18 years) in septic shock and admitted to ICU will be included in the study. Patients will be randomized as per computer generated random number into the Drug (Atorvastatin, 40 mg) or matched placebo group. Drug or placebo will be given to selected patient via nasogastric tube for 7 days. Bio markers (Il-6, TNF-alpha) estimated during the trial week (Days 1, 4, and 7). All clinical and study personnel and patients remained blinded to the study group assignment throughout the trial.

DETAILED DESCRIPTION:
Objectives:

* Study impact of statins on levels of biomarkers (IL-6 and TNF-α) of sepsis.
* Study survival benefit of statins in septic shock.

Introduction:

Sepsis is the leading cause of mortality in non-coronary ICUs. Mortality associated with sepsis is still considerably high. Rising economic burden of managing sepsis is a major concern. Statin is an anti-hyperlipidemic drug with pleiotropic effects. It has properties like anti-inflammatory/oxidative, immunomodulatory effects, enhances endothelial function, reduction in blood thrombogenicity, and increased nitric oxide (NO) bioavailability. Available evidence suggests that statins may play a positive role in reduction of mortality in sepsis. However, the multidimensional heterogeneous character of the available studies does not allow drawing firm conclusions about its usefulness in sepsis and septic shock. This randomized, double blinded, placebo controlled trial is an attempt to study the impact of statins on mortality and biomarker levels in septic shock.

Details of material and methods:

Patients >= age 18 yrs meeting the American European consensus conference definition of septic shock will be enrolled into the study. After the written informed consent from the primary decision maker the patients will be randomized into either the drug or placebo group. Each group will either receive Atorvastatin 40mg or a matched placebo for 7 days. IL-6 and TNF alpha levels will be estimated on D1, D4 and D7 of the trial week. Relevant clinical and laboratory (clinical biochemistry, hematological, coagulation parameters, LFT and renal function tests) will be recorded simultaneously. Severity scores, event free days (vasopressor, ventilation, dialysis, transfusion, parenteral nutrition), and mortality after 28 days of inclusion in study will be recorded.

Ethical Issues:

Written informed consent will be taken from either the patient (if possible) or from the primary decision maker related to the patient.

Study population:

A total of 80 patients of septic shock admitted in ICU will be enrolled into this study. Patients either admitted with septic shock or who develop septic shock during their stay in ICU will be eligible for inclusion into the study. The statin and placebo group will have 40 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Clinical disease of septic shock
* Aged eighteen years and above
* Admitted to ICU

Exclusion Criteria:

* Previous statin induced myopathy or hypersensitivity reaction
* Greater than two and half times elevated liver transaminases
* Chronic liver disease
* Pregnant or lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 day of ICU stay
  28 day mortality after inclusion in study.

SECONDARY OUTCOMES:
Cytokines in septic shock | Day 1, 4 and 7 of commencement of trial drug.
  IL-6, TNF-α levels on Day 1, 4 and 7.
Vasopressor free days. | 28 days after commencement of trial drug.
  Vasopressor free days during septic shock.
Ventilation free days. | 28 days after commencement of trial drug.
  Ventilation free days during septic shock.
Renal replacement free days. | 28 days after commencement of trial drug.
  Renal replacement free days during septic shock.
Transfusion free days. | 28 days after commencement of trial drug.
  Transfusion free days during septic shock.
Total parenteral nutrition free days. | 28 days after commencement of trial drug.
  Total parenteral nutrition free days during septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Ratender K Singh, MD., Principal Investigator — Sanjay Gandhi Post Graduate Institute of Medical Sciences
Locations (2):
- India (2):
  - Department of Critical Care Medicine, Lucknow, Uttar Pradesh
  - Department of Immunology, SGPGIMS, Lucknow, Uttar Pradesh

REFERENCES:
- [Derived] Singh RK, Agarwal V, Baronia AK, Kumar S, Poddar B, Azim A. The Effects of Atorvastatin on Inflammatory Responses and Mortality in Septic Shock: A Single-center, Randomized Controlled Trial. Indian J Crit Care Med. 2017 Oct;21(10):646-654. doi: 10.4103/ijccm.IJCCM_474_16. PMID 29142375